CLINICAL TRIAL: NCT02563535
Title: Evaluation of the Use of ACOTEC Drug-Eluting Balloon Litos ® in Below-The-Knee Arteries to Treat Critical Limb Ischemia
Acronym: ACOART-BTK
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ospedale San Donato (Other)
Responsible Party: Principal Investigator, Leonardo Bolognese, MD, MD, Ospedale San Donato
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Arezzo015
Record Dates: First submitted 2015-09-27; First posted 2015-09-30 (Estimated); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Drug-eluting balloon (Experimental): angioplasty with Litos drug-eluting balloon
  Interventions: Device: DEB
- conventional PTA (Active Comparator): angioplasty with conventional balloon
  Interventions: Device: PTA

INTERVENTIONS:
Device: DEB — angioplasty with Litos drug eluting balloon
  Arms: Drug-eluting balloon
Device: PTA — angioplasty with conventional balloon
  Arms: conventional PTA

SUMMARY:
The aim of this study is to evaluate the potential advantage in terms of late lumen loss reduction of Litos drug-eluting balloon vs standard percutaneous transluminal angioplasty in the treatment of below-the-knee disease in patients with critical limb ischemia.

ELIGIBILITY:
Inclusion Criteria:

* age>18 years
* critical limb ischemia (Rutherford class 4-6)
* angiographic stenosis>50% or occlusion of at least one tibial vessel of at least 40mm for which an interventional treatment is scheduled

Exclusion Criteria:

* need for major amputation known before intervention
* allergy to Paclitaxel
* contraindication for combined antiplatelet treatment
* life expectancy <1 year
* hypersensitivity or contraindication to one of the study drugs
* lack of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2015-09; Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Late Lumen Loss (LLL) in the target lesion documented by angiography | 6 months
  Late Lumen Loss (LLL) in the target lesion documented by angiography

SECONDARY OUTCOMES:
Number of events of angiographic occlusive restenosis | 6 months
  number of events of angiographic occlusive restenosis
Number of events of target lesion revascularization (TLR) | 12 months
  number of events of target lesion revascularization

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiovascular Department, Ospedale S.Donato, Arezzo, AR, Italy